CLINICAL TRIAL: NCT03793218
Title: A Comparison of Alar Batten Graft to the Latera Nasal Implant for the Treatment of Nasal Valve Collapse
Brief Title: Alar Batten Graft vs Latera for Nasal Valve Collapse
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution before participants were enrolled.
Sponsor: University of Virginia (Other)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20859
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Nasal Valve Incompetence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Latera Device (Experimental): The LATERA (Spirox Inc., Menlo Park, CA) device, an absorbable nasal implant comprised of a 70:30 blend of poly(L-lactide) and poly(D-lactide), is designed to provide support to the upper and lower lateral cartilages, thereby correcting nasal wall collapse. The implant was first used in the US and cleared by the FDA in 2016. It is designed as a ribbed cylindrical structure with a forked distal end. The implant is delivered endonasally, with a 16-gauge catheter, lateral to the upper and lower lateral cartilages and over the ascending process of the maxilla. The forked end rests on the ascending process of the maxilla and the flexible implant provides support the nasal sidewall soft tissue and cartilage. This non-toxic, biocompatible co-polymer has an extensive use in a variety of medical devices including suture materials and implants. In vivo studies demonstrate the copolymer to reliably decompose over an 18-24 month period.
  Interventions: Device: Latera Device
- Alar Batten Graft (Active Comparator): This study seeks to compare a "gold standard" functional rhinoplasty maneuver, the alar batten graft, to the LATERA implant
  Interventions: Procedure: Alar Batten Graft

INTERVENTIONS:
Device: Latera Device — This study seeks to compare a "gold standard" functional rhinoplasty maneuver, the alar batten graft, to the LATERA implant
  Arms: Latera Device
Procedure: Alar Batten Graft — This study seeks to compare a "gold standard" functional rhinoplasty maneuver, the alar batten graft, to the LATERA implant
  Arms: Alar Batten Graft

SUMMARY:
Nasal obstruction is a common complaint for the patient presenting to the Otolaryngologist and/or the Facial Plastic surgeon. There are numerous potential causes of nasal obstruction, with more easily addressed pathologies such as posterior septal deviation and inferior turbinate hypertrophy often being over-diagnosed. Nasal valve obstruction, particularly dynamic nasal sidewall collapse, is of significant interest to the rhinoplasty surgeon. Traditionally, collapse of the nasal sidewall has been addressed via structural cartilage grafting, with alar batten grafting being the most commonly used method to provide support to the weak nasal sidewall. Recently, an absorbable nasal implant, comprised of a polylactic acid copolymer, has been advocated for supporting the nasal sidewall and relieving nasal obstruction. There are several proposed advantages of the implant over traditional operative techniques, namely the ease of endonasal insertion, which can be performed in the outpatient clinic setting. Preliminary investigations demonstrate subjective improvement in nasal obstruction with use of the implant, however, there has been no direct comparison with traditional techniques utilizing cartilage grafting.

This study is being done at both UVa and in Oregon. This prospective study will randomize patients with nasal obstruction and documented dynamic nasal sidewall collapse into one of two groups undergoing treatment with either endonasal batten grafting or the absorbable Latera nasal valve implant. Preoperative and postoperative nasal obstruction will be assessed with a validated survey for nasal obstructive symptoms, the Nasal Obstruction Symptom Evaluation (NOSE) score. The mean preoperative and postoperative NOSE score between the groups will be compared at 1, 6, 12, and 24 months post-operatively to compare the efficacy of both techniques. Subjects will be blinded to the surgical intervention they receive.

ELIGIBILITY:
Inclusion Criteria:

* Documented physical exam findings of septal deviation
* Bilateral nasal sidewall collapse on inspiration
* Subjective improvement in nasal obstruction with use of the modified Cottle maneuver

Exclusion Criteria:

* Prior septorhinoplasty
* Obvious trauma to the nose causing nasal obstruction
* Inflammatory conditions such as chronic rhinosinusitis with nasal polyposis
* Patients using chronic topical nasal decongestants or illicit intranasal drug use
* Prisoners, cognitively impaired, non-English speaking subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
12 Month NOSE Score | 12 months
  Mean change in Nose score at 12 month post-op visit

SECONDARY OUTCOMES:
1 Month NOSE Score | 1 month
  Mean change in Nose score at 1 month post-op visit
6 Month NOSE Score | 6 months
  Mean change in Nose score at 6 month post-op visit
24 Month NOSE Score | 24 months
  Mean change in Nose score at 24 month post-op visit